CLINICAL TRIAL: NCT02247219
Title: Promoting Health in Healthy Living Centres - Does it Work, How Does it Work and Why?
Brief Title: Promoting Health in Healthy Living Centres - a Clinical Study Among Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: University of Agder (Other)
Responsible Party: Principal Investigator, Eivind Meland, Professor at the Department of Global Publ Health and Prim Care, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 228454/DHE
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Health Behavior
Keywords: Health education; Health services research
MeSH Terms: conditions — Health Behavior; Health Education | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 'Counselling and education individually and in groups'
  Interventions: Behavioral: Counselling and education individually and in groups
- Waiting list control (Other): The waiting list group waits 6 months after assessment and allocation and is reassessed after 6 and 12 months. Both groups are reassessed after 24 months, and the second part of the study is a one group longitudinal cohort study.
  Interventions: Behavioral: Counselling and education individually and in groups

INTERVENTIONS:
Behavioral: Counselling and education individually and in groups — The counselling method is based om Motivational Interviewing

SUMMARY:
The study aims at:

Using Intervention mapping as a planning approach for behavior change intervention programs, based on an ecological approach to health and local community and user participation.

* Explore the behavioral change processes utilizing qualitative methods.
* Develop theory-based behavior change programs across different domain at healthy living centres.
* Evaluate the effect of behavior change intervention programs across different domains.
* Increase health providers' competence in effective behavioral change intervention techniques by networks and education seminars between municipalities and research groups.
* The programs will specifically target the underlying causes of chronic disease. The investigators will map the distribution of lifestyle habits among individuals and families. The investigators will also explore how lifestyle habits relate to known determinants of social health inequality, such as adverse previous experiences, participation in working life and low income.
* The investigators also intend to study if socioeconomic differences are of importance for entering or dropping out of HLC interventions, and the ability to sustain lifestyle changes. The investigators will do so by stratified analyses, or by using socioeconomic variables as determinants in effect analyses.

DETAILED DESCRIPTION:
Approaches, hypotheses and choice of method

A multidisciplinary team of researchers will work to realize this project according to a systematic stepwise approach that combines the use of the PRECEDE-PROCEED model and Intervention Mapping (IM) protocol. The PRECEDE-PROCEED model is a conceptual model serving the needs of the current project with an educational and ecological approach in health program planning. IM will be used as a planning approach to develop theory- and evidence based health promoting intervention programs. Following the IM process, it maps the path from needs assessment, development of program objectives, selection of intervention methods and strategies, and program design. A benefit of IM is its linkage with community-based participatory research as it includes engagement of community members to identify and refine priority areas. Thus, the process of including IM in developing intervention programs will secure that users and staff in the healthy living centres will have significant autonomy and may influence the development of the intervention programme, and tailor the intervention to fit local needs.

In the initial steps of the IM process will explore the research field utilizing qualitative research methods. The investigators will use focus groups and in-depth interviews to obtain sufficient information to tailor the intervention to local needs and resources. The investigators intend to explore the expectations staff and users of HLCs have about the different intervention programmes, and how they perceive attendance.

The research program will have Self Determination Theory (SDT) as a theoretical point of departure and as an overall theoretical framework for qualitative studies and RCTs of behavioral intervention programs across different behavioural domains. Even though our logic model for understanding behavioral change is linear, focusing on the presumed cause-effect identified in theory and empirical research, the investigators acknowledge that the behavioral treatment programs and proposed outcomes are part of a complex multilevel system (an ecological approach) (Bartholomew et al.2011). An ecological way of analyzing health problems and solutions support the use of a variety of theories when developing a program, as opposed to one single theory. Theories can help in describing the at-risk groups and environmental agents, understand the health-promotion behaviors and environmental agents, understanding the heath-promotion behaviors, and finding methods to promote change (Bartholomew, 2011).

The 0-hypothesis in the controlled studies is that the different behavioral treatment programs have no effects compared with controls. Alternative research hypotheses are:

* Participants who perceive the interpersonal health care-climate as autonomy supportive, will report more autonomous reasons for attending the program and following it's guidelines (self-determined).
* The program will predict increases in autonomous motivation for behavioral change, perceived self-efficacy for program constructs: e.g. physical exercise, healthy eating, and quality of life.
* The program will improve the participants' health behavior.
* The program will improve the participants' self-perceived health and risk factors of non-communicable diseases.

The investigators will also measure effects on health behaviour and health in ordinary practice in the municipalities, in studying effects of systemic and organisational interventions. This will benefit the external validity of the research project.

ELIGIBILITY:
Inclusion Criteria: All persons attending a participating Healthy living center who understands norwegian and can answer the questionnaires -

Exclusion Criteria: Do not understand written norwegian language

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Physical activity changes measured with accelerometer | 6 months
Dietary changes measured with validated questionnaire | 6 months

SECONDARY OUTCOMES:
Wellbeing, self-rated health and body satisfaction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gro B Samdal, Masters, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Undecided
We will share data with faculty members at UoB and UoA based on agreements of analysing and Publishing.

REFERENCES:
- [Derived] Abildsnes E, Meland E, Mildestvedt T, Stea TH, Berntsen S, Samdal GB. The Norwegian Healthy Life Study: protocol for a pragmatic RCT with longitudinal follow-up on physical activity and diet for adults. BMC Public Health. 2017 Jan 5;17(1):18. doi: 10.1186/s12889-016-3981-1. PMID 28056906
- [Derived] Stea TH, Haugen T, Berntsen S, Guttormsen V, Overby NC, Haraldstad K, Meland E, Abildsnes E. Using the Intervention Mapping protocol to develop a family-based intervention for improving lifestyle habits among overweight and obese children: study protocol for a quasi-experimental trial. BMC Public Health. 2016 Oct 18;16(1):1092. doi: 10.1186/s12889-016-3766-6. PMID 27756346
- See also: Home page of principal investigator — http://www.uib.no/personer/Eivind.Meland